CLINICAL TRIAL: NCT04957537
Title: Evaluation of the Effect of a Semantic Rehabilitation in Patients in the Mild to Moderate Stage of Primary Progressive Semantic Aphasia : a SCED Study
Brief Title: Semantic Rehabilitation for Patients With Primary Progressive Semantic Aphasia
Acronym: SCED-APPvs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/21/0215
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Primary Progressive Aphasia
Keywords: Semantic primary progressive aphasia; semantic variant (svPPA); speech therapy; anomia; metacognition; Single Case Experimental Design; technology; naming; speed of lexical access
MeSH Terms: conditions — Aphasia, Primary Progressive; Pick Disease of the Brain; Communication Disorders; Anomia

STUDY DESIGN:
Intervention Model Description: Interventional, monocentric, prospective, randomised, controlled research. Single Case Experimental Design" type study in multiple baselines with 2 successive phases (A-B design) for each patient. For each subject, phase A constitutes the baseline (6 to 8 weeks), phase B is characterised by semantic rehabilitation (5 weeks). The beginning of the intervention will be sequential and the duration of the baseline will be randomised for each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 weeks phase A (Other): According to SCED methodology design :
  Phase A, which constitutes the control period of semantic therapy, will be composed of lexico-phonological training exercises (Piroux-Davous, 2018). This phase will last 6 weeks (i.e. 18 sessions), at the rate of 3 speech therapy sessions of 45 minutes per week.
  Interventions: Behavioral: semantic therapy and semantic re-education
- 8 weeks phase A (Other): According to SCED methodology design :
  Phase A, which constitutes the control period of semantic therapy, will be composed of lexico-phonological training exercises (Piroux-Davous, 2018). This phase will last 8 weeks (i.e. 24 sessions), at the rate of 3 speech therapy sessions of 45 minutes per week.
  Interventions: Behavioral: semantic therapy and semantic re-education

INTERVENTIONS:
Behavioral: semantic therapy and semantic re-education — Patients will be followed over two periods "Phase A (randomized, 6 to 8 weeks) - Phase B (5 weeks)".
  Phase A : Baseline Phase A, which constitutes the control period of semantic therapy, will be composed of lexico-phonological training exercises (Piroux-Davous, 2018). This phase will last 6 to 8 weeks (i.e. 18 to 24 sessions) depending on the randomisation, at the rate of 3 speech therapy sessions of 45 minutes per week.
  Phase B : Semantic re-education The sessions will consist of training based on the analysis of semantic traits (Coustaut, 2019). This phase will last 5 weeks (i.e. 15 sessions), at the rate of 3 speech therapy sessions of 45 minutes per week.
  In accordance with the application of the SCED methodology, repeated measurements will be carried out every second session during phases A and B. They will consist of proposing the oral naming task (lasting 10 minutes).

SUMMARY:
This project aims to measure the effect of a semantic rehabilitation protocol for patients with primary progressive semantic aphasia and using the SCED methodology.

DETAILED DESCRIPTION:
The damage on the semantic system is at the heart of the clinical picture of semantic primary progressive aphasia (PPA), a neuro-evolutionary pathology. In other words, patients gradually lose access to concepts, general knowledge, word memory and meaning. In the absence of effective pharmacological treatment to reduce the symptoms evoked by patients and improve their quality of life, the arguments in favour of speech and language therapy are multiplying.

Numerous lexico-semantic multimodal indication therapies have been described in scientific studies. The most studied is semantic rehabilitation through the analysis of semantic features, which has shown its effectiveness in the context of vascular and post-traumatic aphasia.

However, there are only few studies and applications in neuro-evolutionary pathologies such as semantic PPA and those studies are complicated by methodological biases. It has been shown that relearned knowledge is more likely to be retained and transferred to everyday life (generalisation) if the material used is specific to the needs of each individual. Given the heterogeneity of clinical profiles in neuro-evolving pathologies and the inter-individual variability, the personalised approach should be favoured.

To evaluate the effect of semantic therapy in patients with semantic PPA, this study therefore proposes to use the SCED (Single Case Experimental Design) methodology. In addition to allowing an individual analysis, this methodology has the advantage of corresponding to a high level of evidence due to the acquisition of repeated measures and the randomisation of the introduction of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of primary progressive semantic aphasia according to the criteria of Gorno-Tempini et al (2011) (Appendix A)
* Being in the mild to moderate stage of dementia (MMSE score between 10 and 28) (Crum et al., 1993; Derouesné et al., 1999)
* Common French
* Being affiliated to a social security scheme
* Being over the age of 18 years old

Exclusion Criteria:

* Have significant uncorrected visual and/or hearing impairment
* Have a history of brain injuries, major head trauma
* Have untreated psychiatric disorders
* Have significant motor and/or comprehension problems that make it impossible to take part in the study
* Chronical use of drugs and/or alcohol
* Under guardians or curators
* Severe depression (Beck's depression scale score > 9) (Beck & al., 1961)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Performance in speaking | Baseline (before phase A)
  To evaluate speaking accuracy, the study team will assess the number of correct items recovered by the patient when performing a specific naming task before the rehabilitation.
  The naming task is a selection of 80 items developped by Coustaut in 2019 in its MetaLex protocol.
Performance in speaking | Baseline (before phase A)
  To evaluate speaking response time, the study team will assess the rate at which items are recovered by the patient when performing a specific naming task before the rehabilitation.
  The naming task is a selection of 80 items developped by Coustaut in 2019 in its MetaLex protocol.
Performance in speaking | immediately after the intervention (after phase B)
  To evaluate speaking accuracy, the study team will assess the number of correct items repeated by the patient when performing a specific naming task after the rehabilitation.
  The naming task is a selection of 80 items developped by Coustaut in 2019 in its MetaLex protocol.
Performance in speaking | immediately after the intervention (after phase B)
  To evaluate speaking response time, the study team will assess the rate at which items are recovered by the patient when performing a specific naming task after rehabilitation.
  The naming task is a selection of 80 items developped by Coustaut in 2019 in its MetaLex protocol.

SECONDARY OUTCOMES:
Maintenance of the performance in speaking | 1 month after the end of the intervention (after phase B)
  Number of correct items recovered by the patient when performing a specific naming task 1 month after the end of the intervention.
  The naming task is a selection of 80 items developped by Coustaut in 2019 in its MetaLex protocol.
  This will be compared to the number of items correctly recovered at the end of the rehabilitation (corresponding to outcome 3 here).

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie PARIENTE, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No